CLINICAL TRIAL: NCT06141720
Title: Feasibility of a Mindfulness Intervention for Endometriosis Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Christa Coleman, Assistant Professor, Psychiatry and Behavioral Health, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23397
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis; Pain; Mindfulness
MeSH Terms: conditions — Endometriosis; Pain | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care for endometriosis surgery plus education (Active Comparator)
  Interventions: Behavioral: pain education
- Standard of care for endometriosis surgery plus mindfulness (Experimental)
  Interventions: Behavioral: mindfulness of pain introduction and intervention

INTERVENTIONS:
Behavioral: pain education — Pain education
  Arms: Standard of care for endometriosis surgery plus education
Behavioral: mindfulness of pain introduction and intervention — Brief mindfulness of pain introduction and intervention
  Arms: Standard of care for endometriosis surgery plus mindfulness

SUMMARY:
Endometriosis is a common cause of pelvic pain in women which has been historically under-studied and under-diagnosed. The goal of this research is to pilot-test the feasibility and acceptability of a manualized, single-session brief mindfulness-based intervention (BMBI) among participants with endometriosis-related chronic pelvic pain (ECPP) who undergo surgical treatment, and gather preliminary data necessary for future studies assessing BMBI's impact on outcomes in surgically-treated ECPP. This pilot study will enroll 10-20 adult participants with ECPP to receive either a BMBI adjunctive to treatment as usual (TAU; n=5-10) or education with TAU (n=5-10) prior to their ECPP surgery. The central hypothesis is the BMBI is feasible to deliver pre-operatively, acceptable to patients, and may help improve acute post-surgical outcomes through more adaptive stress coping and pain processing, enabled by mindfulness training.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older
2. diagnosis or probable diagnosis of endometriosis
3. candidate for surgical procedure for endometriosis
4. English speaking
5. have access to wifi and email

Exclusion Criteria:

1. prior formal mindfulness training
2. Unable to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Use of opioid medication | 1 week
  Morphine milligram equivalent following surgery
Use of opioid medication | 3 months
  Morphine milligram equivalent following surgery
Pain intensity | 1 week
  Numerical Pain Rating Scale 0-10, 10 being highest
Pain intensity | 3 months
  Numerical Pain Rating Scale 0-10, 10 being highest

SECONDARY OUTCOMES:
Sleep quality (sleep duration, awakenings, efficiency) | 1 week prior to surgery
  actigraphy monitoring
Sleep quality (sleep duration, awakenings, efficiency) | 1 week following surgery
  actigraphy monitoring
Sleep report | 1 week following surgery
  sleep diary (hours slept, activities during day and night)
Sleep report | 1 week prior to surgery
  sleep diary (hours slept, activities during day and night)
Emotional functioning | baseline
  Hospital Anxiety and Depression Scale 0-21, 21 is worst
Emotional functioning | 1 week
  Hospital Anxiety and Depression Scale 0-21, 21 is worst
Emotional functioning | 3 months
  Hospital Anxiety and Depression Scale 0-21, 21 is worst
Patient global impression of change | 3 months
  Global Impression of change 1-7, 1 is best
Patient global impression of change | 1 week
  Global Impression of change 1-7, 1 is best
Pain catastrophizing | baseline
  Pain catastrophizing Scale 0-52, 52 is worst
Pain catastrophizing | 1 week
  Pain catastrophizing Scale 0-52, 52 is worst
Pain catastrophizing | 3 months
  Pain catastrophizing Scale 0-52, 52 is worst
Treatment satisfaction | 1 week
  Treatment satisfaction 0-10, 10 being best
Treatment satisfaction | 3 months
  Treatment satisfaction 0-10, 10 being best
Heart rate variability | baseline
  brief HRV assessment baseline and during intervention

OTHER OUTCOMES:
Pain threshold | baseline
  Pain threshold
Temporal summation | baseline
  Temporal summation of pain

CONTACTS AND LOCATIONS:
Overall Officials: Christa Coleman, Principal Investigator — Penn State Health
Locations (1):
- Penn State Health, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No